CLINICAL TRIAL: NCT05091177
Title: Study on Correlation Between Cytomegalovirus and Ocular Myasthenia Gravis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: XiaoYong Liu (Other)
Responsible Party: Sponsor-Investigator, XiaoYong Liu, Deputy chief physician, First Affiliated Hospital of Jinan University
Organization: First Affiliated Hospital of Jinan University (Other)
Other Study IDs: 2021JiNan
Record Dates: First submitted 2021-10-09; First posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Ocular Myasthenia Gravis; Cytomegalovirus Infections
MeSH Terms: conditions — Myasthenia Gravis; Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the patience group: underwent the following examinations: serum acetylcholine receptor antibody, erythrocyte deposition rate, hypersensitive C protein, neostigmine test, chest CT, low frequency repetitive nerve stimulation (orbicularis oculi muscle, levator palpebrae muscle, frontalis muscle), thyroid function and color ultrasound.
  Interventions: Diagnostic Test: Serum acetylcholine receptor antibody, erythrocyte deposition rate, hypersensitive C protein, neostigmine test,thymus CT, low frequency repeated nerve stimulation
- the normal group: underwent the following examinations: serum acetylcholine receptor antibody, erythrocyte deposition rate, hypersensitive C protein, neostigmine test, chest CT, low frequency repetitive nerve stimulation (orbicularis oculi muscle, levator palpebrae muscle, frontalis muscle), thyroid function and ultrasound.
  Interventions: Diagnostic Test: Serum acetylcholine receptor antibody, erythrocyte deposition rate, hypersensitive C protein, neostigmine test,thymus CT, low frequency repeated nerve stimulation

INTERVENTIONS:
Diagnostic Test: Serum acetylcholine receptor antibody, erythrocyte deposition rate, hypersensitive C protein, neostigmine test,thymus CT, low frequency repeated nerve stimulation — Use relevant instruments for inspection

SUMMARY:
Ocular myasthenia gravis (OMG) is an autoimmune neuromuscular disease mediated by pathogenic autoantibodies. Its etiology and pathogenesis are not completely clear. The occurrence and development of OMG are the result of the joint participation of genetic factors, environmental factors and immune factors. The role of infectious factors in the pathogenesis of autoimmune diseases is a hot topic in the international discussion.By analyzing the difference in the positive rate and titer of CMV antibodies between ocular myasthenia gravis and healthy people. By analyzing the correlation between the positive rate and titer of CMV antibodies and ocular myasthenia gravis clinical manifestations, acetylcholine receptor antibodies, ESR, hypersensitive C-reactive protein, complement C3, complement C4 and thymus status.To investigate the correlation between cytomegalovirus and ocular myasthenia gravis. It can provide new insights for further studies on the etiology and possible pathogenesis of ocular myasthenia gravis.

DETAILED DESCRIPTION:
A total of 75 patients and 40 healthy volunteers are collected who are diagnosed with ocular myasthenia gravis in the First Affiliated Hospital of Jinan University from January 2019 to January 2022 . All subjects undergo eye examination and cytomegalovirus antibody detection. OMG patients undergo the following examinations: serum acetylcholine receptor antibody, erythrocyte deposition rate, hypersensitive C protein, neostigmine test, chest CT, low frequency repetitive nerve stimulation (orbicularis oculi, levator palpebrae superioris, frontalis muscle), thyroid function and color ultrasound. The difference of lgG positive rate ,lgM positive rate of CMV and antibody titers of lgG and lgM are analyzed between the two groups, and the relationship between CMV antibody and OMG clinical manifestations, acetylcholine receptor antibody, laboratory indicators and thymus status are analyzed.

ELIGIBILITY:
the patience group Inclusion criteria:

* Clinical manifestations: fluctuating eye muscle weakness;
* Positive ice test, fatigue test, rest and sleep test;
* Positive neostigmine test;
* Serum acetylcholine receptor antibody and other antibodies are positive;
* Repeated electrical nerve stimulation test attenuation is positive;
* Meeting the above diagnostic criteria of the first, or any of the other 4, at the same time excluding other diseases caused by eye palsy can be clear diagnosis.

the patience group exclusion criteria:

* General myasthenia gravis;
* History of other eye diseases
* With other autoimmune diseases or other inflammatory diseases;
* Patients with diabetes, hypertension, coronary heart disease and other chronic medical history or cancer diseases;
* Hepatitis B virus, hepatitis C virus, HIV, syphilis positive patients;
* immunosuppressive drugs (such as glucocorticoid, azathioprine and cyclosporine A), gamma globulin for intravenous injection, plasmapheresis, etc., within 3 months before treatment;
* Previous thymic resection or thymus radiation therapy;
* Pregnancy or lactation.

the control group Inclusion criteria:

* No obvious abnormality was found in the recent physical examination results;
* No history of autoimmune diseases;
* Have not received antiviral therapy or immunotherapy within 3 months;
* No history of other eye diseases or systemic diseases.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of 75 patients and 40 healthy volunteers are collected who are diagnosed with ocular myasthenia gravis in the First Affiliated Hospital of Jinan University from January 2019 to January 2022
Sampling Method: Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
CMV lgG, lgM positive rate | 1year
  CMV-lgG titer ≥14IU/ mL is positive, 12-14 IU/ mL is critical, and 0-12 IU/ mL is negative. CMV-lgM titer > 22U/ mL is positive, 18-22U/mL is critical, and 0-18U/mL is negative.
CMV lgG, lgM antibody titer | 1year
  Concentrations of cytomegalovirus lgG and lgM antibodies is collected for analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided